CLINICAL TRIAL: NCT03272945
Title: Linked-color Imaging Versus White Light for the Detection of Colorectal Flat Lesions: a Randomized, Controlled Trial
Brief Title: Linked-color Imaging for the Detection of Colorectal Flat Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief of Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: LCI
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCI (Experimental): Once the randomization assignment was announced, the whole colonoscopy from insertion to cecum to withdrawal of endoscope was carried out entirely by using Linked-color imaging (LCI).
  Interventions: Procedure: Linked-color imaging
- WL (Placebo Comparator): Once the randomization assignment was announced, the whole colonoscopy from insertion to cecum to withdrawal of endoscope was carried out entirely by using white light (WL).
  Interventions: Procedure: Linked-color imaging

INTERVENTIONS:
Procedure: Linked-color imaging — Linked-color imaging colonoscopy

SUMMARY:
Linked color imaging (LCI) was recently developed and uses a laser endoscopic system (Fujifilm Co, Tokyo, Japan) that acquires images by simultaneously using narrow-band short-wavelength light and white-light (WL) in an appropriate balance. LCI is a new image-enhancing technology that is intended to enhance slight color differences in the red region of the mucosa. The acquired color information is reallocated to differentiate colors that are similar to the mucosal color, resulting in improved performance in depicting blood vessels, and additional image processing that enhances color separation for red color permits clear visualization of red blood vessels and white pits. This modality may increase the detection rate of colorectal polyps by enhancing the visibility of colonic mucosal vessels. In addition, it has been reported that LCI increases the visibility of colorectal flat lesions and contributes to improvement of the detection rate for these lesions. The primary aim of the current study was to compare the detection rate of colorectal flat lesions of LCI cap-assisted colonoscopy with WL cap-assisted colonoscopy in prospective randomized trial. In addition, we prospectively compared LCI and WL with regard to the visibility of colorectal flat lesions found in this study.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled consecutive patients who were referred for colonoscopy to our hospital for diagnostic work up of colonic symptoms, surveillance of colorectal polyps, and colorectal cancer screening.

Exclusion Criteria:

* familial colorectal cancer syndrome including familial adenomatous polyposis and hereditary non-polyposis colorectal cancer syndrome, personal history of colorectal cancer or inflammatory bowel disease and those who had previous colonic resection.

Patients who were considered to be unsafe for polypectomy, including patients with bleeding tendency and those with severe comorbid illnesses, were excluded. Those in whom <90% of mucosa was seen due to mixture of semisolid and solid colonic contents were also excluded because of poor bowel preparation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Average prevalence of flat lesion /patient detected | procedure
  The total number of flat colorectal lesion/patient was defined. The average prevalence of flat lesion /patient detected was calculated.

SECONDARY OUTCOMES:
Adenoma detection rate | procedure
  Adenoma detection rate was defined as the proportion of patients with at least one adenoma found on colonoscopy.
Polyp detection rate | procedure
  Polyp detection rate was defined as the proportion of patients with at least one polyp found on colonoscopy.

OTHER OUTCOMES:
The visibility of colorectal flat lesions | 1 day
  Six endoscopists interpreted the images of CLI and WL. By using a previously reported visibility scale, we scored the visibility level on a scale of 1 to 4 and compared the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, MD, Principal Investigator — Showa Inan General Hospital
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kudo T, Horiuchi A, Kyodo R, Horiuchi I, Arai N, Kajiyama M, Tanaka N. Linked colour imaging versus white-light colonoscopy for the detection of flat colorectal lesions: A randomized controlled trial. Colorectal Dis. 2021 Jun;23(6):1414-1420. doi: 10.1111/codi.15605. Epub 2021 Mar 16. PMID 33645911